CLINICAL TRIAL: NCT00722436
Title: Tranexamic Acid for the Reduction of Allogeneic Blood Exposure in Infants and Children Having Craniofacial Surgery
Brief Title: Tranexamic Acid for Craniofacial Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study dose changed based on recent publications
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Franklyn Cladis, Associate Professor of Anesthesiology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO07120134
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Craniosynostosis; Bleeding
Keywords: antifibrinolytic, tranexamic acid
MeSH Terms: conditions — Craniosynostoses; Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic acid (Experimental): Tranexamic acid (100 mg/kg load, 10 mg/kg/hr) intravenous
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): Saline was administered intravenously
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Tranexamic acid — 100 mg/kg load, then 10 mg/kg/hr
  Arms: Tranexamic acid
Drug: saline — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, blinded, prospective study that will investigate the potential benefit of tranexamic acid to reduce the intraoperative bleeding and blood transfusions in pediatric patients undergoing craniofacial surgeries.

DETAILED DESCRIPTION:
Surgical procedures for the correction of craniofacial deformities result in unavoidable and significant blood loss in small children and infants. Patients may experience blood losses that exceed one to two blood volumes. In an effort to reduce our transfusion requirements, we have introduced tranexamic acid into our practice. However, the benefit of tranexamic acid in pediatric craniofacial surgery has not yet been reported. We hypothesize that the intraoperative use of tranexamic acid in pediatric patients presenting for craniofacial reconstructions will reduce blood loss and allogeneic transfusion requirements.

This is a randomized, blinded, prospective study that will investigate the potential benefit of tranexamic acid to reduce the intraoperative bleeding and blood transfusions in pediatric patients undergoing craniofacial surgeries. An initial dose of 100 mg/kg tranexamic acid (Cyclokapron 100mg/ml) or an equal volume of a placebo will be administered over 15 minutes after the induction of anesthesia and before the skin incision. A maintenance infusion of 10 mg/kg/hr of tranexamic acid or equal volume of a placebo will be started upon completion of the initial dose and will be continued until skin closure. The primary outcome will include the reduction in the total volume of allogeneic erythrocytes.

ELIGIBILITY:
Inclusion Criteria:

The inclusion of the patients will depend on the following criteria:

1. All pediatric patients scheduled for primary or secondary repair of craniosynostosis with a frontal orbital advancement, or cranial vault reconstruction.
2. Patients will be between the ages of 6 months and 18 years old.
3. They will be > than 5 kg.
4. All subjects being evaluated in the Craniofacial Clinic for primary or secondary repair of craniosynostosis will potentially be included in the study. Prior to inclusion in the study potential participants will be screened by history and laboratory data. The laboratory data will include a complete blood count, PT, PTT, type and cross, factor V leiden, anticardiolipin antibody, and lupus anticoagulant. The history will be obtained from the parents or current care takers. The medical records may be reviewed if there is a need for clarification.

Exclusion Criteria:

Patients that will be excluded from the study include the following:

1. Familial or personal coagulopathy risk-factor V leiden, anticardiolipin antibody, and lupus anticoagulant
2. Abnormal PT, PTT, Platelet count. or closing time. All patients presenting for craniofacial surgery have preoperative blood work performed which includes a type and screen, HCT, PLT, PT, PTT, and closing time. Patients who have abnormalities detected in their coagulation profile proceed on to a complete hematologic evaluation that includes an evaluation for Von Willebrand's Disease.
3. History of thrombotic episodes in the patient
4. Renal failure or hepatic failure.
5. Infants less than 5 kg
6. Age < 6 months or > 18 years old

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We stopped the study early because emerging data came out that demonstrated benefit with significantly lower doses than our study. We were compelled to stop enrolling.

REFERENCES:
- [Background] Neilipovitz DT, Murto K, Hall L, Barrowman NJ, Splinter WM. A randomized trial of tranexamic acid to reduce blood transfusion for scoliosis surgery. Anesth Analg. 2001 Jul;93(1):82-7. doi: 10.1097/00000539-200107000-00018. PMID 11429344
- [Background] Sethna NF, Zurakowski D, Brustowicz RM, Bacsik J, Sullivan LJ, Shapiro F. Tranexamic acid reduces intraoperative blood loss in pediatric patients undergoing scoliosis surgery. Anesthesiology. 2005 Apr;102(4):727-32. doi: 10.1097/00000542-200504000-00006. PMID 15791100
- [Background] Henry DA, Moxey AJ, Carless PA, O'Connell D, McClelland B, Henderson KM, Sly K, Laupacis A, Fergusson D. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2001;(1):CD001886. doi: 10.1002/14651858.CD001886. PMID 11279735

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranexamic Acid: Tranexamic acid (100 mg/kg load, 10 mg/kg/hr)
  Tranexamic acid: 100 mg/kg load, then 10 mg/kg/hr
  Patients are randomized to TXA or saline. This group is the TXA group.
- Placebo: Saline
  saline: Placebo
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 11 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Total Volume (ml/kg) of Allogeneic Blood Exposure.
Description: This is the blood administered during surgery. The blood comes form the blood bank. It is not cell salvage blood. The volume was normalized by weight.
Time Frame: intraoperative and postoperative (24 hr)
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 9 | 11
ml/kg | 16.1 (13.9) | 17.1 (10.4)

2. Primary Outcome: Number of Patients That Remained Transfusion Free
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 9 | 11
participants | 2 | 0

3. Secondary Outcome: Effect of Tranexamic Acid on Prothrombin Time (PT), Partial Thromboplastin Time (PTT) at Three Time Points (Baseline, After Osteotomies, and Immediately After Procedure).
Time Frame: (baseline, after osteotomies, and immediately after procedure)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 9 | 11
seconds
  PT -baseline | 15.1 (0.84) | 13.8 (0.74)
  PT-after osteotomies | 18.5 (3.93) | 16.1 (1.94)
  PT-immediately after surgery | 17.7 (1.18) | 17 (1.74)
  PTT -baseline | 34.6 (2.92) | 32.9 (2.67)
  PTT-after osteotomies | 37.2 (9.75) | 34.6 (3.62)
  PTT-immediately after surgery | 33.3 (3.5) | 34.8 (3.9)

4. Secondary Outcome: Platelets
Time Frame: baseline, after osteotomies, immediately after surgery
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 9 | 11
10^9 platelets/L
  platelets-baseline | 301 (109) | 364 (125)
  platelets-after osteotomies | 253 (101) | 300 (107)
  platelets-immediately after surgery | 223 (89) | 231 (99)

ADVERSE EVENTS:
Arm/Group | Tranexamic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

LIMITATIONS AND CAVEATS:
Study terminated because two studies published during the trial demonstrated efficacy of tranexamic acid at a lower dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes